CLINICAL TRIAL: NCT02609295
Title: Effects of α-linolenic Acid Supplementation in the Form of Perilla Oil on Collagen-epinephrine Closure Time, Activated Partial Thromboplastin Time and Lp-PLA2 Activities in Nondiabetic and Hypercholesterolemic Subjects
Brief Title: Effects of α-linolenic Acid Supplementation on Hemostasis in Nondiabetic and Hypercholesterolemic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HP-ALA-hyperchol
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Hypercholesterolemia
Keywords: α-linolenic acid; perilla oil; aPTT; Collagen-epinephrine closure time; Lp-PLA2
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Individuals who consumed 1.2 g (two capsules) of medium-chain triglyceride (MCT) oil daily
  Interventions: Dietary Supplement: Placebo
- ALA group (Experimental): Individuals who consumed 1.2 g (two capsules) of perilla oil daily
  Interventions: Dietary Supplement: ALA group

INTERVENTIONS:
Dietary Supplement: Placebo — 1.2 g (two capsules) of medium-chain triglyceride (MCT) oil
  Arms: Placebo
Dietary Supplement: ALA group — 1.2 g (two capsules) of perilla oil
  Arms: ALA group

SUMMARY:
This study evaluates whether ALA intake alters total cholesterol and homeostatic factors and the relationship between these alteration and lipoprotein associated phospholipase A2 (Lp-PLA2) activity.

DETAILED DESCRIPTION:
An 8-week, randomized, double-blind, placebo-controlled study was conducted with 86 nondiabetic and borderline-to-moderate hypercholesterolemic (200mg/dL ≤ serum cholesterol ≤ 300mg/dL) subjects, not taking any medications and supplements to affect lipid metabolism, platelet function and inflammation, divided into two groups: an α-linolenic acid (ALA) group [1.2 g (two capsules) of perilla oil daily; 497 mg ALA] and a placebo group (1.2 g of medium-chain triglyceride oil daily).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate and sign in informed consent form
* Adults aged 40-70
* Nondiabetic and hypercholesterolemic subjects (serum cholesterol ≥ 200 mg/dL)

Exclusion Criteria:

* Subjects taking any medication or supplements known to affect lipid metabolism or platelet function, n-3 fatty acid supplementation or n-3 fatty acid-rich fish more than two times per week
* Following diseases: dyslipidemia, hypertension, diabetes, liver disease, renal disease, pancreatitis, cardiovascular disease, gastrointestinal disease, cancer, or any other disease requiring treatment
* Participation in clinical trials of any drug or supplement within 30 days prior to the participation of the study
* Pregnant or lactating women, alcoholic, mental patient
* Judged to be inappropriate for the study by the investigator after reviewing other reasons

Ages: 40 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Collagen-Epinephrine Closure Time (C-EPI CT) | Baseline
Collagen-Epinephrine Closure Time (C-EPI CT) | 8-week follow up

SECONDARY OUTCOMES:
Prothrombin Time (PT) | Baseline
Prothrombin Time (PT) | 8-week follow up
Activated partial thromboplastin time (aPTT) | Baseline
Activated partial thromboplastin time (aPTT) | 8-week follow up
Fibrinogen | Baseline
Fibrinogen | 8-week follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University, Seoul, South Korea